CLINICAL TRIAL: NCT01507623
Title: The Role of Capnography in Endoscopy Patients Undergoing Nurse Administered Propofol Sedation (NAPS): A Randomized Study
Brief Title: Value of Capnography During Nurse Administered Propofol Sedation (NAPS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Collaborators: The Ministry of Science, Technology and Innovation, Denmark (Other Government)
Responsible Party: Principal Investigator, Charlotte Slagelse, Medical Student, University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NAPS_CAPNOGRAPHY1
Record Dates: First submitted 2011-11-24; First posted 2012-01-11 (Estimated); Last update posted 2012-01-11 (Estimated); Status verified 2012-01

CONDITIONS: Hypoxia
Keywords: NAPS; Hypoxia; Propofol; capnography; endoscopy; Sedation
MeSH Terms: conditions — Hypoxia | interventions — Capnography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- With Capnograpy (Experimental): Intervention group with the addition of capnography to standard monitoring (non-invasive blood pressure, pulse, pulse oximetry, clinical observation of respiration, electrocardiography (ECG) and respiratory frequency measured by the ECG)
  Interventions: Device: Capnography (Phillips MP20 monitor)
- No Capnography (No Intervention): Control group without the addition of capnography to standard monitoring (non-invasive blood pressure, pulse, pulse oximetry, clinical observation of respiration, electrocardiography (ECG) and respiratory frequency measured by the ECG)

INTERVENTIONS:
Device: Capnography (Phillips MP20 monitor) — In the intervention group the NAPS nurse observed possible hypoxia and changes in capnography curves/values during the procedure and was instructed to decrease propofol and take actions against insufficient ventilation* if etCO2 ≥ 7kPa or ≤ 2 kPa for ≥ 1 minute, if respiratory frequency ≤ 8 or a loss of curve shape was registered.
  *Suction, increase oxygen supply, tongue holder or nasal airway, bag-mask ventilation,paged anaesthesia Discontinued procedures
  Other Names: Capnography: Phillips MP20 monitor; Nasal cannulae: Smart CapnoLine GuardianTM
  Arms: With Capnograpy

SUMMARY:
Propofol is widely used by anaesthesiologists for deep sedation and general anaesthesia. During recent years nurses trained in the use of low dose Propofol sedation (NAPS) during endoscopy have been introduced. The method has been implemented at the endoscopic unit at Gentofte hospital since 2008(1). Propofol has a respiratory depressive effect which may result in depressed oxygen saturation in the blood (hypoxia). Due to a short acting half life this is prevented in the majority of cases. However, in spite of this, hypoxia is experienced in 4,4% of patients receiving propofol during endoscopy at Gentofte Hospital (unpublished data). It is well known that hypoxia constitutes a late expression of reduced oxygen tension in peripheral tissues. Whether the addition of capnography to standard monitoring during NAPS may be of benefit is widely unknown. The aim of this study is to examine whether the additional use of capnography to standard monitoring during endoscopy may improve patient safety in patients undergoing low dose Propofol sedation by reducing the number, duration and level of hypoxic events. The trial is a randomized clinical prospective case-control study.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 or above
* compliant with the criteria of NAPS.

Exclusion Criteria:

* no signed written consent obtained
* American Society of Anaesthesiologists (ASA) physical status classification > 3
* sleep apnoea
* allergy against soy, eggs and peanuts
* body Mass Index (BMI) > 35 kg/m2
* mallampati Score ≥ 4
* acute gastrointestinal bleeding
* subileus
* ventricular retention
* severe COLD ((30% ≤ FEV1 <50%)
* failed data collection

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 591 (Actual)
Dates: Start 2010-09; Primary Completion 2011-02 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
The number of hypoxic events | The sum of events registered during procedures (procedure duration is, depending on the type, 3 to 90 minutes)
  If the addition of capnography to standard monitoring can reduce the number of hypoxic events in patients undergoing endscopy with NAPS. A hypoxic event is defined as an observed oxygen saturation of less than 92% . Data is collected by a computer with intervals of 12 sec as the smallest possible.

SECONDARY OUTCOMES:
Actions taken against respiratory insufficiency | Registered during procedure(procedure duration is, depending on the type, 3 to 90 minutes)
  Whether more or less actions are taken against respiratory insufficiency with or without capnography in patients undergoing endoscopy with NAPS.
The duration of hypoxia | The sum of time with hypoxia registered during procedures (procedure duration is, depending on the type, 3 to 90 minutes)
  The duration of hypoxia is measured as the sum of registrations(each registration represents 12 seconds) with an oxygen saturation of less than 92 percent. Data is collected by a computer with intervals of 12 sec as the smallest possible.
The level of hypoxia | The sum of events registered at each level during procedures (procedure duration is, depending on the type, 3 to 90 minutes)
  Saturation is registered every 12 seconds into a computer. Hypoxia (saturation <92%) was divided into three levels of hypoxia: 1. <92% - 90%,2. <90% - 88%, 3. <88%.
  And the number of events in each group was summed up.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Vilmann, MD, Prof., Study Director — Herlev and Gentofte University Hospital, Denmark; Charlotte Slagelse, Med. student, Principal Investigator — Gentofte University Hospital, Denmark
Locations (1):
- Gentofte University Hospital, Hellerup, Denmark

REFERENCES:
- [Derived] Slagelse C, Vilmann P, Hornslet P, Jorgensen HL, Horsted TI. The role of capnography in endoscopy patients undergoing nurse-administered propofol sedation: a randomized study. Scand J Gastroenterol. 2013 Oct;48(10):1222-30. doi: 10.3109/00365521.2013.830327. Epub 2013 Sep 2. PMID 23992025